CLINICAL TRIAL: NCT03128970
Title: Synchronizing Blastocyst at Hatching Stage in Frozen Embryo Transfer Cycles
Brief Title: Synchronizing Blastocyst in Frozen Embryo Transfer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Yasmeen Fertility and Gynecology Center (Other)
Collaborators: Ganna Fertility Center (Other)
Responsible Party: Principal Investigator, Yasmin Magdi, Dr, Al-Yasmeen Fertility and Gynecology Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 001-2017
Record Dates: First submitted 2017-04-21; First posted 2017-04-25 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Embryo Implantation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The gynecologist performing the embryo transfer as well as the patients undergoing frozen embryo transfer will be blinded to group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- frozen/thawed (No Intervention): blastocysts with three or less grade of expansion will be thawed and then subsequently transferred into women uterus three hours post-thawing.
- synchronized frozen/thawed hatching blastocysts (Experimental): blastocyst thawing (with three or less grade of expansion) will take place the day before embryo transfer in order to reach hatching stage
  Interventions: Other: synchronizing blastocysts

INTERVENTIONS:
Other: synchronizing blastocysts — transferring frozen/thawed a synchronized blastocysts at hatching stage into female uterus.
  Arms: synchronized frozen/thawed hatching blastocysts

SUMMARY:
The aim of the present study is to determine if implantation rate could be increased in women undergoing frozen embryo transfer cycles in case of adjusting their embryo development at hatching stage.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who will agree to participate and assign an informed consent form
2. Only blastocyst transfer FET cycles
3. Patients undergoing FET after their 1st IVF or ICSI cycle with no pregnancy at the fresh transfer
4. Freeze-all cycles due to OHSS
5. Freeze-all cycles due to poor endometrium
6. Age 19-33 at the time of randomization.
7. Their frozen blastocysts are 3 or less grade of expansion.
8. Female with a ≥12 AFCs
9. Endometrial thickness ≥ 8mm at the time of ovulation
10. Women with their male partners will give only fresh semen
11. Women who have no uterine abnormality by ultrasound
12. BMI ≤ 31

Exclusion Criteria:

1. Cycles undergoing preimplantation genetic diagnosis.
2. Women who have previous two cycles of implantation failure at fresh transfer
3. Women who have previous two FET failed cycles
4. Any uterine pathology (myomas, adenomyosis, endocrinopathies, thrombophilia, chronic pathologies, acquired or congenital uterine abnormalities)
5. Patients with severe endometriosis
6. Presence of uni- or bilateral hydrosalpinx
7. Recurrent pregnancy loss.
8. Any medical condition that affect fertility.

Ages: 19 Years to 33 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 742 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
Ongoing implantation rate | 12 weeks
  ultrasound detection of ongoing gestational sacs with heartbeats after 12 weeks of gestation per transferred embryos

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Al-Yasmeen fertility and gynecology center, Banhā
  - Ganna Fertility and Gynecology Center, Cairo

IPD SHARING:
Plan to Share IPD: Yes